CLINICAL TRIAL: NCT00225290
Title: Double-blind, Placebo-controlled, Randomized Phase III Trial of Oral Thalidomide in Advanced Hepatocellular Carcinoma With Poor Liver Reserve
Brief Title: Phase III Trial of Oral Thalidomide in Advanced Hepatocellular Carcinoma With Poor Liver Reserve
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slowly recruitment rate
Sponsor: TTY Biopharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T2202
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2005-09

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Phase III; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

INTERVENTIONS:
Drug: Thalidomide(Thado)

SUMMARY:
To compare the overall survival of thalidomide- and placebo-treated advanced HCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with measurable, metastatic or locally advanced hepatocellular carcinoma
2. The diagnosis of HCC should be established either by cyto/histology
3. Patients must be > 20 years of age.
4. ECOG score < 2.
5. Signed informed consent.
6. Female patients at child-bearing age must have negative pregnancy test.

Exclusion Criteria:

1. Patients with other systemic diseases which require concurrent usage of glucocorticosteroid or immunosuppressant agent(s) are not eligible.
2. Patients with advanced second primary malignancy are not eligible.
3. Patients with active infection are not eligible.
4. Patients with pregnancy or breast-feeding are not eligible.
5. Patients with brain metastases are not eligible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2003-02

PRIMARY OUTCOMES:
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, M.D Ph.D., Principal Investigator — Division of Cancer Research, National Health Research Institute Ward 191
Locations (1):
- Taiwan Cooperative Oncology Group, Taipei, Taiwan